Reflow Medical Wingman Catheter Wing-IT Clinical Trial RFM-CTO-13001 NCT03403426

Document Date: 03-OCT-2018

## PROTOCOL SUMMARY

Title: A Non-Randomized Study Evaluating the Use of the ReFlow Medical

Wingman Catheter to Cross Chronic Total Occlusions in Infrainguinal

Peripheral ArTeries (Wing-IT)

Design: Prospective, multi-center, non-randomized single-arm study of the

> Wingman Catheter to cross a single infrainguinal peripheral chronic total occlusion (CTO). Safety and effectiveness will be evaluated during the

index procedure through 30-day follow-up.

To evaluate the safety and effectiveness of the ReFlow Medical **Purpose:** 

Wingman Catheter used to cross de novo or restenotic infrainguinal

CTOs that cannot be crossed with a standard guidewire.

**Enrollment** and A maximum of 85 patients will be enrolled and treated with the

Sites: investigational device at up to twelve (12) centers in North America and

three (3) centers in Europe.

**Time Course:** Initial enrollment: O1 2018

> Last enrollment: O1 2019 Last follow-up: Q1 2019

**Primary Efficacy and** Primary Efficacy:

**Safety Endpoints:** While using the Wingman device, successful CTO crossing is identified by successful guidewire placement in the distal true lumen confirmed by

angiography with no clinically significant perforations.

Primary Safety:

No evidence of significant in-hospital or 30-day MAEs. No evidence of clinically significant perforation, clinically significant embolization or ≥

Grade C dissection, after Wingman CTO crossing and prior to

adjunctive interventions, confirmed by angiography. Components of the

composite primary safety endpoint include:

Major Adverse Events (MAEs) defined as death, unplanned target limb major amputation, and emergent target vessel revascularization.

- Clinically significant perforation defined as all perforations requiring intervention (e.g., covered stent, bypass or other surgery) 1
- Clinically significant embolization defined as those events that result in distal ischemia (e.g., occlusion of run-off vessel

- resulting in pain or foot discoloration) and/or requires rescue intervention.
- Grade C Dissection or greater with a minimum of a dissection protruding outside the lumen of the vessel persisting after passage of the contrast material.<sup>1</sup>

The components of the primary and secondary safety endpoints will be adjudicated by an independent CEC with angiographic elements assessed by an independent core laboratory.

## **Secondary Endpoints:**

- 1) Lesion success, defined as attainment of <50% final residual stenosis of the target lesion using any percutaneous method.
- Procedure success, defined as device success and the absence of inhospital MAEs, clinically significant perforation, clinically significant embolization or Grade C or greater dissection not resolved by visual estimate.
- 3) Procedure safety, defined as any in-hospital AE or MAE following use of a therapeutic interventional device.
- 4) Evaluation of total procedural and fluoroscopic time and contrast volume.
- 5) Evaluation of procedure time associated with use of the investigational device.
- 6) Evaluation of utility of ancillary device in addition to investigational device.

## **Inclusion Criteria:**

- 1) Patient is willing and able to provide informed consent.
- 2) Patient is willing and able to comply with the study protocol.
- 3) Patient is > 18 years old.
- 4) Patient has peripheral arterial disease requiring revascularization as evidenced by contrast, CT or MR angiography.
- 5) Patient has at least one but not more than two occluded infrainguinal arteries that are 99-100% stenosed and no flow is observed in the distal lesion except the flow from collateral circulation.
- 6) Target lesion(s) is  $\geq 1$  cm and < 30 cm in length by visual estimate.
- 7) Target vessel is  $\geq 2.0$  mm in diameter.
- 8) Patient has Rutherford Classification of 2-5.
- 9) Lesion cannot be crossed by concurrent conventional guidewire.
- 10) Reconstitution of vessel at least 2cm above bifurcation/trifurcation.
- 11) Occlusion can be within previously implanted stent.

## **Exclusion Criteria:**

- 1) Patient has a known sensitivity or allergy to contrast materials that cannot be adequately pre-treated.
- 2) Patient has a known sensitivity or allergy to all anti-platelet medications.
- 3) Patient is pregnant or lactating.
- 4) Patient has a co-existing disease or medical condition contraindicating percutaneous intervention.
- 5) Target lesion is in a bypass graft.

- 6) Patient has had a failed crossing attempt without an intervening intervention on the target limb within the past 14 days.
- 7) Patient has a planned surgical or interventional procedure within 30 days after the study procedure.

**Data Analysis** Syntactx

4 World Trade Center Center:

150 Greenwich Street / 44th Floor

New York, NY 10007

**Sponsor:** ReFlow Medical, Inc.

1003 Calle Sombra,

San Clemente, CA 92673

**Principal** 

**Investigator:** Dr. John Laird

**Angiographic Core** 

Yale Cardiovascular Research Group Lab

135 College Street, Suite 101

New Haven, CT 06510